CLINICAL TRIAL: NCT01619124
Title: Part I: Incidence, Clinical Course and Significance of MRI for Early Diagnosis of Osteonecrosis in Children and Adolescents With Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma (LBL) Part II: Susceptibility for Aseptic Osteonecroses in Children and Adolescents With Chemotherapy for ALL or LBL
Brief Title: Osteonecroses in Pediatric Patients With ALL
Acronym: OPAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinik für Kinder-Onkologie, -Hämatologie und Klinische Immu (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kinder-Onkologie, -Hämatologie und Klinische Immu, principal investigator and senior physician university paediatric clinic, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: DKS 2011.11
Record Dates: First submitted 2012-06-06; First posted 2012-06-14 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Osteonecrosis; Acute Lymphoblastic Leukaemia; Lymphoblastic Lymphoma
Keywords: osteonecrosis; children; pediatric; acute lymphoblastic leukaemia; lymphoblastic lymphoma
MeSH Terms: conditions — Osteonecrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Nowadays approximately 80% of children and adolescents with acute lymphoblastic leukaemia (ALL) or lymphoblastic lymphoma (LBL) can be cured and become long-term survivors. Avascular osteonecroses (ON) appear as serious side-effect of antileukaemic treatment. Frequently ON are first diagnosed at higher and than irreversible stages (ARCO III, IV). At these advanced stages curative treatment options are not available. Hence ON are associated with considerable morbidity concerning pain and immobility and go along with long-term impairment of quality of life. Therefore early diagnosis of ON in the follow-up of children and young adults with ALL or LBL is a pressing object.

Within the prospective multicentric observational OPAL-trial patients at risk (aged 10 years or older) treated according to the clinical trials ALL-BFM(Berlin-Frankfurt-Muenster Study Group), COALL or NHL (Non Hodgkin Lymphoma)-BFM in Germany should be examined with regard to the development of ON. By using a treatment associated, risk orientated assessment and examination incidence, symptoms and the clinical course of ON are investigated. The validity of MRI screening in the early diagnosis of ON in children and young adults is analysed.

Systematical investigation of patients under antileukaemic treatment is intended to contribute to risk adapted diagnostic strategies and to serve as data base for the subsequent evaluation of preventive and interventional approaches for the treatment of ON. Long-term objective is the reduction of ON-associated morbidity.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ALL or LBL
* age at diagnosis of ALL or LBL ≥ 10 and < 18 years
* study patient of AIEOP( Associazione Italiana Ematologia ed Oncologia Pediatrica)-BFM, COALL or NHL-BFM in Germany
* treatment in a hospital participating in OPAL
* written informed consent

Exclusion Criteria:

* relapse of ALL or LBL
* every non evidence based treatment (pharmacological, orthopaedic-conservative, orthopaedic operative) aiming at the prevention of ON during study participation
* pacemaker, other MRI prohibited devices
* metal implants in the field of view, other MRI prohibited implants
* pregnancy
* claustrophobia

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with acute lymphoblastic leukemia or lymphoblastic lymphoma, aged >= 10 and < 18 years
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
occurence of early ON stages | 6 years
  Calculation of the rate of by MRI detectable (still) asymptomatic patients with early ON stages (I and II) within the patients who develop symptomatic ON in the further course

SECONDARY OUTCOMES:
ON incidence | 6 years
  Prospective evaluation of incidence of asymptomatic and symptomatic ON in children and adolescents with ALL or LBL

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Kuhlen, Dr. med., Study Chair — Heinrich-Heine University, Duesseldorf
Locations (25):
- Germany (25):
  - Department of Paediatric and Adolescend Medicine, University Aachen, Aachen
  - Department of Pediatrics, Haematology and Oncology, University Bonn, Bonn
  - Department for Children and Adolescent Helth Chemnitz gGmbH, Chemnitz
  - Clinic of Pediatric and Adolescent Medicine, Vestische Caritas Clinic Datteln, Datteln
  - Division of Pediatric Hematology and Oncology, University Children´s Hospital, Dresden
  - Clinic of Pediatric Oncology, Hematology and Clinical Immunology, Center for Child and Adolescent Health, Heinrich Heine University, Düsseldorf
  - Clinic of Pediatrics and Adolescent , Pediatric Hematology and Oncology, Erlangen
  - Department of Pediatric-Oncology/-Hematology and clin. Immunology, University Medicine Essen, Essen
  - Department of Pediatric Hematology, Oncology and Hemostaseology, Goethe-University, University Children's Hospital, Frankfurt am Main
  - Pediatric Hematology and Oncology, University Medicine Greifswald, Greifswald
  - Clinic of Pediatric Hematology and Oncology, University Medical Center Hamburg-Eppendorf, Hamburg
  - Department of Pediatric and Adolescent Helth, University Medical Center Heidelberg, Heidelberg
  - Clinic and Polyclinic of Oncology and Haematology, Herdecke, Herdecke
  - Children's Hospital Medical Center, Pediatric Haematology and Oncology, Homburg
  - Clinic of Pediatric Hematology and Oncology, Kassel, Kassel
  - Department of Pediatrics, University Medicine of Schleswig-Holstein, Campus Kiel, Kiel
  - Clinic of Pediatric and Adolescent Helth, Koblenz-Mayen, Koblenz
  - Helios Klinikum Krefeld Department of Paediatric and Adolescent Medicine, Krefeld
  - Clinic of Oncology and Hematology, Johannes Wesling Klinikum, Minden
  - Department of Paediatric Oncology and Hematology, Cnopf'sche Kinderklinik, Neuendettelsau
  - Department of General Pediatrics, Hematology and Oncology Oldenburg gGmbH, Oldenburg
  - Clinic of Paediatric and Adolescend, University Rostock, Rostock
  - Clinic of Paediatric Oncology and Hematology, Helios Klinikum Schwerin, Schwerin
  - Clinic Trier, Klinikum Mutterhaus der Bromäerinnen, Trier
  - Department of Pediatrics and Adolescent Medicine, University Medical Center Ulm, Ulm